CLINICAL TRIAL: NCT06580080
Title: Evaluation of Are You Ready?
Acronym: AYR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Policy & Research Group (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Mathematica Policy Research, Inc. (Other); Reproductive Health National Training Center (Unknown); Institute of Women & Ethnic Studies (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1 TP2AH000094-01-00
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Teen Pregnancy Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Are You Ready? (Experimental)
  Interventions: Behavioral: Are You Ready? (AYR)
- Social Media Awareness Shorts (Sham Comparator)
  Interventions: Behavioral: Social Media Awareness Shorts (SMAS)

INTERVENTIONS:
Behavioral: Are You Ready? (AYR) — AYR is a group-based entertainment education (EE) intervention designed for sexually active youth who are at risk for or involved in the juvenile justice and/or child welfare systems. AYR is delivered in one, 2.5-hour (150-minute) session with a group of between 2 to 20 youth. The session includes screening a 40-minute video, "Happy Birthday, Leonard" and group-based discussions led by one to two facilitators. Discussions are guided by a participant workbook with journal prompts and handouts.
  The session includes two modules; each module involves screening approximately 20 minutes of "Happy Birthday, Leonard" followed by a 40-minute group discussion. Module 1 includes topics related to contraception, condom use (with a condom demonstration), healthy communication, and stress management. Module 2 includes topics related to condom negotiation, communication styles, and intergenerational cycles.
  Arms: Are You Ready?
Behavioral: Social Media Awareness Shorts (SMAS) — SMAS is a virtually delivered, individual-based health program focused on social media use awareness. Participants are directed to a learning management platform that contains a pre-recorded, facilitated program. The program involves watching several short films and independently completing several activities related to social media use. The program does not include information related to the primary outcomes for this study.
  Arms: Social Media Awareness Shorts

SUMMARY:
The goal of this randomized trial is to learn if the Are You Ready? (AYR) intervention has a positive impact on the sexual and mental health behaviors of sexually active youth between the ages of 14 and 21 years old who are at risk for or involved in the juvenile justice and/or child welfare systems. The primary research questions it aims to answer are:

* Three months after being offered the intervention, does AYR impact youth's receipt of sexually transmitted infection testing in the past three months?
* Three months after being offered the intervention, does AYR impact youth's use of coping skills?
* Nine months after being offered the intervention, does AYR impact youth's frequency of having vaginal and anal sex without condoms in the past three months?

Researchers will compare participants randomized to receive AYR (treatment group) to participants randomized to receive a control condition that contains no sexual or reproductive health information (control group).

Participants randomized to the treatment group will be offered AYR as a virtual or in-person, 2.5 hour group session. Participants randomized to the control group will be offered a virtually delivered control condition.

DETAILED DESCRIPTION:
This is an individual-level, randomized control trial to rigorously evaluate the impact of the Are You Ready? (AYR) intervention. Participant outcomes will be assessed using self-reported, individual-level data gathered using a structured questionnaire administered at three time points: baseline (enrollment); three months post-intervention (four months after baseline); and nine months post-intervention (ten months after baseline).

ELIGIBILITY:
Inclusion Criteria:

* At risk for or involved in the juvenile justice and/or child welfare systems
* Has had vaginal or anal sex in the past 6 months
* Comfortable reading, speaking, and writing in English

Exclusion Criteria:

* Has received other known sexual and reproductive health evidence-based interventions implemented in their local area.
* Enrolled in an ongoing PRG-run TPP study
* Identified as fraudulent

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1850 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-09-14 (Estimated)

PRIMARY OUTCOMES:
Receipt of sexually transmitted infection (STI) testing in the past three months | Assessed three months after the intervention period has ended (four months post-baseline)
  Participants are asked the following item:
  1) Have you been tested for sexually transmitted infections (STIs) in the past 3 months? The resulting variable is dichotomous with values 0 or 1, where 0 indicates a person who has not received STI testing in the past three months and 1 indicates a person who has received STI testing in the past three months.
Use of coping skills | Assessed three months after the intervention period has ended (four months post-baseline)
  Participants are asked on a 4-point scale ranging from "I did not use" (1) to "I used almost all the time" (4) how often they used the following strategies:
  1. I talked to someone to find out more about the situation.
  2. I let people know what I needed.
  3. I talked to someone who could act in some way to change the situation.
  4. I asked for ideas from a friend who I could trust.
  5. I made a great effort to make things work.
  6. I spent time with someone I wanted to be with.
  7. I tried to look after my health by eating food that was good for me.
  8. I tried to eat regularly.
  9. I made a plan of action and followed it through.
  10. I tried to release my anger by exercising.
  11. I tried to look after myself by getting plenty of sleep.
  12. I tried to be physically fit. The measure is calculated as the average response to all 12 items in the scale.
Times having vaginal and anal sex without condoms in the past three months | Assessed nine months after the intervention period has ended (ten months post-baseline)
  Participants are asked the following two items:
  1. In the past 3 months, how many times have you had vaginal sex without you or your sexual partner using a condom?
  2. In the past 3 months, how many times have you had anal sex without you or your sexual partner using a condom? The resulting variable is continuous with values that range from 0 to k, where 0 indicates that a person has not engaged in vaginal and anal sex without a condom in the past three months, and k indicates the number of times the person has engaged in vaginal and anal sex without a condom in the past three months.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Walsh, PhD, Principal Investigator — The Policy & Research Group
Locations (1):
- The Policy & Research Group, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
A dataset will be prepared at the conclusion of the study, which includes de-identified individual-level data on all study participants who contributed self-report data. Respondents will be represented only by a research ID number. Included in the dataset will be self-report data collected across all survey administrations (including demographic characteristics, sexual behaviors, and theoretical antecedents to those behaviors) and select information on program participation (e.g., which program components were completed). Basic data cleaning steps will be taken in order to ensure data are unidentifiable and to increase usability.
Supporting Information: SAP
Time Frame: The individual participant dataset will become available twelve months after the study has concluded.